CLINICAL TRIAL: NCT03867695
Title: SERRATHOR Trial : Analgesic Effect of Serratus Plane Block After Video-Assisted Thoracoscopic Surgery Lobectomy
Brief Title: SERRATHOR TRIAL : Interest of the Novel Serratus Plane Block in Post Operative Analgesia After Video-Assisted Thoracoscopic Lobectomy
Acronym: SERRATHOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 6755
Record Dates: First submitted 2019-03-01; First posted 2019-03-08 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-03

CONDITIONS: Video Assisted Thoracoscopic Surgery; Lobectomy; Pain Post Operative; Regional Anesthesia
Keywords: Serratus plane block; Analgesia after VATS; Lobectomy VATS
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Block (Experimental): At the end of the lobectomy VATS procedure, 0,5 mL/kg of 0.375% ropivacaine will be administered.
  Under ultrasonography assistance, block will be performed at the fifth rib in the midaxillary line. Local anesthetic will be injected either superficial to the serratus anterior muscle or deep underneath the muscle.
  Anesthesiologists, and all the nurses and caring staff involved in this study will be blinded. Solutions of ropivacaine will be prepared identically by the central pharmacy, without any possible identification of the product.
  Interventions: Drug: Ropivacaine
- Placebo Block - Control Group (Placebo Comparator): Patients will receive a placebo injection with 0,5 mL/kg of sterile normal solution. Under ultrasonography assistance, placebo will be injected at the fifth rib in the midaxillary line, either superficial to the serratus anterior muscle or deep underneath the muscle.
  Anesthesiologists, and all the nurses and caring staff involved in this study will be blinded. Solutions of sterile saline will be prepared identically by the central pharmacy, without any possible identification of the product.
  Interventions: Drug: sterile saline

INTERVENTIONS:
Drug: Ropivacaine — At the end of the lobectomy VATS procedure, 0,5 mL/kg of 0.375% ropivacaine will be administered.
  Arms: Serratus Block
Drug: sterile saline — Patients will receive a placebo injection with 0,5 mL/kg of sterile normal solution
  Arms: Placebo Block - Control Group

SUMMARY:
Pain after thoracic surgery remains a challenge for anesthetists. Although VATS for lobectomy is associated with fewer complications compared to thoracotomy, pain after VATS needs to be treated with opioids. Opioids may lead to PONV, respiratory depression, sedation and pruritus. As part of multimodal analgesia and opioids sparing, several local regional techniques has been described: paravertebral block, thoracic epidural analgesia, intercostal block. To date, there is no gold standard for regional anesthesia after VATS.

Serratus plane block is a local regional technique, recently described for analgesia after breast surgery and ribs fracture. In our hospital center, since 2016, we used the Serratus plane block for patients scheduled for lobectomy VATS : a local retrospective trial showed that SPB was associated with a lower consumption of morphine.

The purpose of this randomized controlled double blinded study is to evaluate the analgesic effect of the Serratus plane block, added to a general anesthesia on post operative pain control after VATS lobectomy.

ELIGIBILITY:
Inclusion criteria:

* All patients undergoing lobectomy VATS
* Older > 18 years
* Patients who meet criteria of ASA 1 to 3 class

Exclusion criteria:

* Patient's refusal to participate in the study
* Psychiatric disorder (impossibility to collect the informed consent)
* Patient under juridical protection
* On going an other study
* Non balanced epilepsy
* 3 grade auriculo-ventricular heart block without pacing
* Severe hepatocellular insufficiency
* Anti arrhythmic treatment : class III of the Vaughan William's classification
* Pregnant patient or/and breastfeeding
* History of opioid abuse
* Allergy to local anesthetic drug or opioids

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Total intravenous morphine consumption (mg) in the PACU and department. | 24 hours
  Including the dose of titration while the patient is in PACU and PCA up to 24h postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Bob HEGER, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided